CLINICAL TRIAL: NCT00908336
Title: Phase II, Multicenter, Randomized, Open Label Study of a Sequential Treatment of Intermittent Erlotinib and Docetaxel Versus Erlotinib in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer After Failure of a Prior Chemotherapy Regimen
Brief Title: Erlotinib and Docetaxel in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) After Failure of One Chemotherapy Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Vicente Alberola Candel, ASOCIACIÓN TERAPEUTICA EN HEMATOLOGÍA Y ONCOLOGÍA MÉDICAS H. ARNAU DE VILANOVA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25033
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Adenocarcinoma; Carcinoma, Non-Small Cell; Lung Neoplasms; Docetaxel; Erlotinib; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma; Lung Neoplasms | interventions — Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel and Erlotinib (Experimental): Patients in the experimental arm will receive sequential treatment of intermittent erlotinib and docetaxel up to 4 cycles in the absence of disease progression, unacceptable toxicity, patient refusal or investigator's decision to discontinue the treatment.
  After 4 cycles, participants will receive 150 mg of erlotinib per day until disease progression, unacceptable toxicity, patient refusal or investigator's decision to discontinue the treatment.
  Interventions: Drug: Docetaxel and Erlotinib
- Erlotinib (Active Comparator): Erlotinib (Tarceva®) 150 mg/day po daily until disease progression, unacceptable toxicity, patient refusal or investigator's decision to discontinue the treatment.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Docetaxel and Erlotinib — Docetaxel (Taxotere®) 75 mg/m2 iv first day of each 21-day cycle. Erlotinib (Tarceva®) 150 mg po days 2-16 of each 21-day cycle. Total: 4 cycles in the absence of disease progression
  Arms: Docetaxel and Erlotinib
Drug: Erlotinib — 150 mg/day po daily
  Arms: Erlotinib

SUMMARY:
Erlotinib has demonstrated efficacy as a single agent in patients with NSCLC and the addition of erlotinib to chemotherapy has not achieved better results in the general population.

However, several preclinical and phase I studies have shown that a sequential treatment of erlotinib and chemotherapy could avoid a possible negative interaction between both drugs when administrated concomitantly, and therefore, it could improve the benefit of the combination therapy.

This study will investigate if the intermittent treatment of a chemotherapy drug, such as docetaxel, with erlotinib could achieve a clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age >= 18 years.
* Histologically or cytologically documented inoperable, locally advanced (stage IIIb with malignant pleural or pericardial effusion) or metastatic (Stage IV) NSCLC.
* Patients who have failed only one prior chemotherapy to treat the advanced disease and candidates to receive a second line treatment.
* ECOG PS 0-2.
* Adequate hematological function: hemoglobin => 9 g/dl; neutrophils count => 1.5 x 10(9)/l; platelet count => 100 x 10(9)/l.
* Adequate liver function: Bilirubin <= 1,5 x ULN; AST and ALT <= x 3 ULN when no hepatic metastases or <=5 x ULN if hepatic metastases; Alkaline phosphatase <=5 x UNL except that there is hepatic metastases.
* Adequate renal function: Calculated creatinine clearance => 40 mL/min (Cockroft y Gault) or serum creatinine <= 1.5 x ULN .
* Patient able to meet the requirements of the study and accessible for correct follow-up.
* Oral swallowing capability.

Exclusion Criteria:

* Previous treated with more than one chemotherapeutic treatment for NSCLC
* Concomitant treatment with another drug under investigation.
* Pregnancy or lactation. Fertile women must provide a negative result of pregnancy test (in serum or urine) within 7 days prior to study treatment start. In addition, they must use an effective method of contraception (oral contraceptives, intrauterine device, barrier methods of contraception, together with spermicidal jelly or surgical sterilization) during the study.
* Evidence of other disease, metabolic or neurological dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications.
* Contraindication for the use of erlotinib or docetaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients without disease progression after 6 months of treatment. | 6 months

SECONDARY OUTCOMES:
Progression-free survival | Time from randomization until objective tumor progression or death for any cause. Tumour progression will be assessed every 2 months.
Duration of Response | The time from the first complete response or partial response until objective tumor progression or death due to progression disease. Tumour progression will be assessed every 2 months.
Overall Response Rate | The proportion of patients with tumor size reduction (complete response or partial response following RECIST criteria). Response will be assessed every 2 months.
Disease Control Rate | The proportion of patients without tumor size increase (complete response, partial response or stable disease following RECIST criteria). Response wil be assessed every 2 months.
Overall survival | Time from randomization until death from any cause. Follow up wil be assessed every 3 months after finishing study treatment.
Safety profile | Toxicity will be discribed per cycle and per patient according to CTCAE vs. 3, every 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Juan, Doctor, Principal Investigator — Hospital Arnau de Vilanova de Valencia; Gaspar Esquerdo, Doctor, Principal Investigator — Hospital Clínica de Benidorm; Alfredo Sánchez, Doctor, Principal Investigator — Hospital Provincial de Castellón; Sonia Maciá, Doctor, Principal Investigator — Hospital General de Elda; Vicente Giner, Doctor, Principal Investigator — Hospital de Sagunto; José Muñoz, Doctor, Principal Investigator — H. Universitario Dr. Peset; Antonio López, Doctor, Principal Investigator — Hospital San Juan de Alicante; Francisco Aparisi, Doctor, Principal Investigator — Hospital Virgen de los Lirios
Locations (8):
- Spain (8):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital San Juan de Alicante, Alicante, Alicante
  - Hospital Clínica de Benidorm, Benidorm, Alicante
  - Hospital General de Elda, Elda, Alicante
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia